CLINICAL TRIAL: NCT00395915
Title: Randomized Evaluation of the Effectiveness of Clozapine and Aripiprazole Versus Clozapine and Haloperidol in the Treatment of Schizophrenia. An Independent, Pragmatic, Multicentre, Parallel-Group, Superiority Trial.
Brief Title: Randomized Evaluation of the Effectiveness of Clozapine and Aripiprazole Versus Clozapine and Haloperidol in the Treatment of Schizophrenia
Acronym: CHAT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universita di Verona (Other)
Responsible Party: Corrado Barbui MD, University of Verona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-004708-38
Record Dates: First submitted 2006-11-03; First posted 2006-11-06 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Schizophrenia
Keywords: schizophrenia; antipsychotics; treatment non response; pragmatic trial
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: aripiprazole

SUMMARY:
The principal clinical question to be answered by CHAT (Clozapine Haloperidol Aripiprazole Trial) is the relative efficacy and tolerability of combination treatment with clozapine plus aripiprazole compared to combination treatment with clozapine plus haloperidol in patients with an incomplete response to treatment with clozapine over an appropriate period of time.

ELIGIBILITY:
Inclusion Criteria:

1. Current treatment with clozapine for the primary indication of schizophrenia (clinical diagnosis, guided by DSM-IV criteria).
2. Treatment with clozapine for at least six months at a stable dose of 400 mg or more per day, unless the size of the dose was limited by side-effects.
3. Unsatisfactory benefit from clozapine treatment, as indicated by the presence of positive symptoms (delusions, hallucinations, abnormal behaviour, clinical diagnosis)
4. Age 18 and above.
5. Agreement between investigator and patient to enter the study.
6. The patient is normally resident in Italy.
7. It is considered clinically reasonable to try combination treatment with clozapine and aripiprazole or with clozapine and haloperidol.
8. Uncertainty about which trial treatment would be best for the participant.
9. No medical disorder or condition contraindicates either of the investigational drugs.
10. Agreement between investigator and patient to discontinue any antipsychotic drugs other than clozapine (including long-acting antipsychotic drugs).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2006-09; Primary Completion 2009-03 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Withdrawal from allocated treatment within 3 months.

SECONDARY OUTCOMES:
Withdrawal from allocated treatment within 12 months of follow-up.
Time to withdrawal from allocated treatment.
Severity of illness, measured at month 3 and 12.
Withdrawal from study treatment, due to adverse reactions, within 3 and 12 months.
Concurrent use of adjunctive medication within 3 and 12 months.
Concurrent use of antiparkinson medication within 3 and 12 months.
Adverse events within 3 and 12 months.
Biological parameters, measured at month 3 and 12.
Metabolic syndrome within 3 and 12 months.
Subjective tolerability of antipsychotic drugs, measured at month 3 and 12.
Deliberate self-harm within 3 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Tansella, MD, Study Chair — Universita di Verona
Locations (1):
- University of Verona, Verona, Italy

REFERENCES:
- [Derived] Cipriani A, Accordini S, Nose M, Purgato M, Girlanda F, Tansella M, Barbui C. Aripiprazole versus haloperidol in combination with clozapine for treatment-resistant schizophrenia: a 12-month, randomized, naturalistic trial. J Clin Psychopharmacol. 2013 Aug;33(4):533-7. doi: 10.1097/JCP.0b013e318296884f. PMID 23775051
- [Derived] Barbui C, Accordini S, Nose M, Stroup S, Purgato M, Girlanda F, Esposito E, Veronese A, Tansella M, Cipriani A; CHAT (Clozapine Haloperidol Aripiprazole Trial) Study Group. Aripiprazole versus haloperidol in combination with clozapine for treatment-resistant schizophrenia in routine clinical care: a randomized, controlled trial. J Clin Psychopharmacol. 2011 Jun;31(3):266-73. doi: 10.1097/JCP.0b013e318219cba3. PMID 21508849
- [Derived] Nose M, Accordini S, Artioli P, Barale F, Barbui C, Beneduce R, Berardi D, Bertolazzi G, Biancosino B, Bisogno A, Bivi R, Bogetto F, Boso M, Bozzani A, Bucolo P, Casale M, Cascone L, Ciammella L, Cicolini A, Cipresso G, Cipriani A, Colombo P, Dal Santo B, De Francesco M, Di Lorenzo G, Di Munzio W, Ducci G, Erlicher A, Esposito E, Ferrannini L, Ferrato F, Ferro A, Fragomeno N, Parise VF, Frova M, Gardellin F, Garzotto N, Giambartolomei A, Giupponi G, Grassi L, Grazian N, Grecu L, Guerrini G, Laddomada F, Lazzarin E, Lintas C, Malchiodi F, Malvini L, Marchiaro L, Marsilio A, Mauri MC, Mautone A, Menchetti M, Migliorini G, Mollica M, Moretti D, Mule S, Nicholau S, Nose F, Occhionero G, Pacilli AM, Pecchioli S, Percudani M, Piantato E, Piazza C, Pontarollo F, Pycha R, Quartesan R, Rillosi L, Risso F, Rizzo R, Rocca P, Roma S, Rossattini M, Rossi G, Rossi G, Sala A, Santilli C, Sarao G, Sarnicola A, Sartore F, Scarone S, Sciarma T, Siracusano A, Strizzolo S, Tansella M, Targa G, Tasser A, Tomasi R, Travaglini R, Veronese A, Ziero S. Rationale and design of an independent randomised controlled trial evaluating the effectiveness of aripiprazole or haloperidol in combination with clozapine for treatment-resistant schizophrenia. Trials. 2009 May 15;10:31. doi: 10.1186/1745-6215-10-31. PMID 19445659